CLINICAL TRIAL: NCT05369559
Title: Mini Bolus for Fluid Challenge Responsiveness in the Emergency Department
Acronym: MIBORED
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Head chief, Emmergency Department ,University Hospital of Monastir, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TN2020-NA T -INS-399
Record Dates: First submitted 2022-03-14; First posted 2022-05-11 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Fluid Therapy

STUDY DESIGN:
Intervention Model Description: The fluid challenge is given intravenously via a specific venous line.
  Patients are assigned in a random chronological order to:
  * receive a "mini-bolus ":50 ml of crystalloid solution, regularly infused over 30 seconds
  * and passive leg raising.
  Passive leg raising technique: Initially, the patient is placed semi-recumbent with the head of the bed at 45°. After recording baseline measurement, the head of the bed is lowered and the legs are elevated to 45° for 2 minutes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mini Bolus 50 (Active Comparator): receiving a "mini-bolus A":50 ml of crystalloid solution, regularly infused over 30 seconds
  Interventions: Diagnostic Test: passive leg rising test
- PLR (Other): Passive leg raising technique: Initially, the patient is placed semi-recumbent with the head of the bed at 45°. After recording baseline measurement, the head of the bed is lowered and the legs are elevated to 45° for 2 minutes
  Interventions: Combination Product: Mini bolus 50

INTERVENTIONS:
Combination Product: Mini bolus 50 — receiving a "mini-bolus A":50 ml of crystalloid solution, regularly infused over 30 seconds
  Arms: PLR
Diagnostic Test: passive leg rising test — Passive leg raising technique: Initially, the patient is placed semi-recumbent with the head of the bed at 45°. After recording baseline measurement, the head of the bed is lowered and the legs are elevated to 45° for 2 minutes
  Arms: Mini Bolus 50

SUMMARY:
Intravascular volume expansion is a common intervention in critically ill patients with acute circulatory failure.we test the hypothesis that a mini-bolus fluid challenge, of either 50 ml , can predict fluid responsiveness in spontaneously breathing patients with hemodynamic instability.

DETAILED DESCRIPTION:
Background:

Intravascular volume expansion is a common intervention in critically ill patients with acute circulatory failure. Nevertheless, approximately 50% of critically ill patients will not benefit from an intravascular volume expansion, since they are in the horizontal portion of the Frank-Starling curve.

Thus, an accurate assessment of fluid responsiveness prior to volume expansion is mandatory to avoid fluid overload, which has been associated with increased morbidity and mortality in critically ill patients.

Fluid challenge, which consists of administering fluid to assess volume responsiveness, is widely performed. However, repeated fluid challenges, several times a day, can be harmful Indeed, if cardiopulmonary function cannot compensate for the increase in preload, fluid loading can compromise micro-vascular perfusion and oxygen delivery or aggravate peripheral and pulmonary oedema.

For many years, spontaneous breathing was considered a major limitation to assess fluid responsiveness in critically ill patients .

In this study, the investigator test the hypothesis that a mini-bolus fluid challenge of 50 ml can predict fluid responsiveness in spontaneously breathing patients with hemodynamic instability.

Passive leg raising technique: Initially, the patient is placed semi-recumbent with the head of the bed at 45°. After recording baseline measurement, the head of the bed is lowered and the legs are elevated to 45° for 2 minutes.

Fluid challenge responsiveness:

Fluid responsiveness is defined as an increase in the cardiac output measured using FloTrac-Vigileo monitor (∆CO-PLR > 10%) after the PLR, separating the studied population into responders and non-responders.

Measurements:

Patients characteristics, including age and sex, are recorded at admission. The aetiology of acute circulatory failure, the inotropic and/or vasopressor support (epinephrine, norepinephrine and dobutamine) and the APACHE II score are recorded.

The following hemodynamic variables are recorded: heart rate (beats per minute), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and mean arterial blood pressure (mmHg). These variables are collected at baseline (T0), immediately before mini-bolus infusion (T50b, T50a), and immediately before the PLR manoeuvre (TPLRb and TPLRa).

Cardiac output (CO) and stroke volume (SV) are measured using both an EsCCO monitor (COescco and SVescco) and a FloTrac transducer connected to a Vigileo monitor (COflotrac and SVflotrac). CO and SV are measured at baseline, before and after each mini-bolus infusion, and before and after passive leg raising. They are recorded at the moment when they plateau. The hemodynamic variables cited above are also recorded at that time.

Changes -induced by the mini-boluses and by the PLR- in all parameters were measured; these were referred to as ∆[parameter]50 and ∆[parameter]PLR.

If patients were treated with norepinephrine, the dose remained unchanged from before volume expansion until all hemodynamic measurements were complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous breathing
* Patients in whom a fluid challenge is indicated because they present acute circulatory failure (which is defined as systolic blood pressure less than 90 mmHg or the need for vasopressors (norepinephrine more than 0.1 µg/kg/min) to maintain a systolic blood pressure more than 90 mmHg (14), and at least one sign of inadequate tissue perfusion:

  * urine output of below 0.5ml/kg per hour over 1 hour
  * tachycardia (heart rate of greater than 100 beats per minute)
  * mottled skin.
  * lactate > 2 mmol/l

Exclusion Criteria:

* Cardiac arrest
* Acute respiratory distress syndrome
* Coma Glasgow Scale < 14
* Age of less than 18 years
* Moribund patients
* Pregnant patients
* impossibility to perform passive leg raising (PLR) (trauma patients, lower extremity amputees, and prone patients)
* Patients with cardiac arrhythmias
* Patients with cardiogenic pulmonary oedema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-08-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Measurement of the cardiac flow with the Estimate Continuous CO escco and SVescco (EsCCO) to predict the fluid responsiveness . | at 3 minutes following fluid load in the day of admission
  Predicting fluid responsiveness in spontaneously breathing patients with hemodynamic instability.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Prof, Principal Investigator — University Hospital Fattouma Bourguiba Monastir , Emergency Department .
Locations (2):
- Tunisia (2):
  - Emergency Departement, Monastir
  - Emergency department, Monastir